CLINICAL TRIAL: NCT03678532
Title: Effects of Sedation on Clinical, Gasometric and Respiratory Muscle Parameters in Critically Ill COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Associate Professor of Anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sedation in COPD
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Sedation in Critically Ill COPD Patients
Keywords: sedation; COPD; critically ill; intensive care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Critical Illness | interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily interruption of sedation (control group) (Experimental): Control group received daily interruption of sedation. After intubation, patients received IV infusion of midazolam. 1-2 mg / hour with increments 1-2 mg/hr gradually increasing dose till RASS reached -4 or -5. Infusion stopped at 7:00 AM. If the patient is awake no need for resuming infusion. If signs of discomfort occurred, infusion resumed at half of the prior dose, targeting conscious sedation (RASS 0: -3)
  Interventions: Drug: Midazolam
- No sedation (Experimental): Intervention group were managed by no-sedation strategy. Patients received bolus doses of midazolam (1-5 mg) only when needed, after atrial to control agitation by correcting the underlying cause. If the patient needed more than 3 bolus doses , IV infusion of midazolam was given by the daily interruption protocol as in the control group. No crossover was allowed between groups. Analysis was done by intension-to-treat principle.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam

SUMMARY:
the investigators conducted a randomized controlled trial in respiratory intensive care unit (RICU) of Assiut University Hospital. COPD patients admitted to RICU were included. Exclusion criteria include: Marked renal impairment, Liver cell failure, neurological disorders, age <18 or >70 and pregnancy.

Patients were randomly allocated to two groups. Midazolam was used for sedation in both groups. Richmond agitation-sedation score (RASS) was used to monitor level of sedation or agitation. Control group received daily interruption of sedation. intervention group managed by no-sedation strategy.

Primary outcome measure: changes in PaCO2 Secondary outcome measures include: changes in PH, heart rate, mean arterial blood pressure, respiratory rate, P0.1 and NIF.

DETAILED DESCRIPTION:
The researchers conducted a randomized controlled trial in respiratory intensive care unit (RICU) of Assiut University Hospital. COPD patients admitted to RICU were included. Exclusion Criteria include: Marked renal impairment (creatinine > 2mg/dl), Liver cell failure (Bilirubin> 3mg/dl), neurological disorders, age <18 or >70 and pregnancy.

Patients were randomly allocated to two groups. Midazolam was used for sedation in both groups. Richmond agitation-sedation score (RASS) was used to monitor level of sedation or agitation. Control group received daily interruption of sedation. After intubation, patients received IV infusion of midazolam, gradually increasing dose till RASS reached -4 or -5. Infusion stopped at 7:00 AM. If the patient is awake no need for resuming infusion. If signs of discomfort occurred, infusion resumed at half of the prior dose, targeting conscious sedation (RASS 0: -3) Intervention group were managed by no-sedation strategy. Patients received bolus doses of midazolam only when needed, after atrial to control agitation by correcting the underlying cause. If the patient needed more than 3 bolus doses , IV infusion of midazolam was given by the daily interruption protocol as in the control group. No crossover was allowed between groups. Analysis was done by intension-to-treat principle.

Follow up arterial blood gas sampling was done baseline at intubation. 1hr., 2hrs., 12hrs., 24hrs. and 48hrs. after intubation. Recording of clinical monitoring parameters (hear rate, mean arterial blood pressure, respiratory rate) was done at the same intervals. Airway occlusion pressure (P0.1) and negative inspiratory force (NIF) were measured 48 hours after intubation to test affection of respiratory muscles in both groups.

Primary outcome measure: changes in PaCO2 Secondary outcome measures include: changes in PH, heart rate, mean arterial blood pressure, respiratory rate, P0.1 and NIF.

ELIGIBILITY:
Inclusion Criteria:

Critically ill patients diagnosed as COPD, admitted to the respiratory intensive care unit (RICU) of Assiut University Hospital.

Exclusion Criteria:

Marked renal impairment (creatinine > 2mg/dl), Liver cell failure (Bilirubin> 3mg/dl), neurological disorders, age <18 or >70 and pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
ventilation affection | 48 hours
  changes in PaCO2 measured in mmHG

SECONDARY OUTCOMES:
effect of sedation on acid base status | 48 hours
  changes in PH
Effect of sedation on heart rate | 48 hours
  heart rate beat per minute changes
Effect of sedation on blood pressure | 48 hours
  including mean arterial blood pressure in mmHg

REFERENCES:
- [Background] Laerkner E, Stroem T, Toft P. No-sedation during mechanical ventilation: impact on patient's consciousness, nursing workload and costs. Nurs Crit Care. 2016 Jan;21(1):28-35. doi: 10.1111/nicc.12161. Epub 2015 Apr 17. PMID 25892407
- [Background] Toft P, Olsen HT, Jorgensen HK, Strom T, Nibro HL, Oxlund J, Wian KA, Ytrebo LM, Kroken BA, Chew M. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation (NONSEDA Trial): study protocol for a randomised controlled trial. Trials. 2014 Dec 20;15:499. doi: 10.1186/1745-6215-15-499. PMID 25528350
- [Background] Strom T, Toft P. Sedation and analgesia in mechanical ventilation. Semin Respir Crit Care Med. 2014 Aug;35(4):441-50. doi: 10.1055/s-0034-1382156. Epub 2014 Aug 11. PMID 25111642
- [Background] Kress JP, Vinayak AG, Levitt J, Schweickert WD, Gehlbach BK, Zimmerman F, Pohlman AS, Hall JB. Daily sedative interruption in mechanically ventilated patients at risk for coronary artery disease. Crit Care Med. 2007 Feb;35(2):365-71. doi: 10.1097/01.CCM.0000254334.46406.B3. PMID 17205005